CLINICAL TRIAL: NCT02317419
Title: PHASE IA/IB, OPEN-LABEL, MULTICENTER, MULTIPLE ASCENDING DOSE STUDY FOLLOWED BY AN EXTENSION PHASE TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND ACTIVITY OF RO6927005, AN ANTI-MESOTHELIN (MSLN) RECOMBINANT CYTOLYTIC FUSION PROTEIN (cFP), ADMINISTERED EITHER ALONE (PART A) OR IN COMBINATION WITH GEMCITABINE AND NAB-PACLITAXEL (PART B) IN PATIENTS WITH MESOTHELIN-POSITIVE METASTATIC AND/OR LOCALLY ADVANCED MALIGNANT SOLID TUMORS
Brief Title: A Study of RO6927005 Either As Monotherapy (Part A) or in Combination With Gemcitabine and Nab-Paclitaxel (Part B) to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Clinical Activity in Patients With Mesothelin-positive Metastatic and/or Locally Advanced Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was prematurely terminated because the emerging benefit:risk ratio did not justify continuing dosing patients.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP29387; 2014-002935-32 (EudraCT Number)
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
Keywords: Solid Cancers
MeSH Terms: conditions — Neoplasms | interventions — LMB-100; Gemcitabine; 130-nm albumin-bound paclitaxel

ARMS (5):
- Part A MAD Phase RO6927005 Monotherapy (Experimental): RO6927005 given as a single agent in participants with tumors known to be mesothelin expressing and with mesothelin-positive tumors. MAD = multiple ascending dose.
  Interventions: Drug: RO6927005
- Part A Extension Phase Group 1 (Experimental): RO6927005 given as a single agent in participants with mesothelin-positive refractory/recurrent solid tumors, other than malignant pleural mesothelioma (MPM) and pancreatic ductal adenocarcinoma (PDA)
  Interventions: Drug: RO6927005
- Part A Extension Phase Group 2 (Experimental): RO6927005 given as a single agent in participants with mesothelin-positive metastatic and/or advanced PDA
  Interventions: Drug: RO6927005
- Part B MAD Phase (Experimental): RO6927005 with gemcitabine/nab-paclitaxel in participants with mesothelin-positive metastatic and/or advanced PDA
  Interventions: Drug: RO6927005; Drug: gemcitabine; Drug: nab-paclitaxel
- Part B Extension Phase (Experimental): RO6927005 with gemcitabine/nab-paclitaxel in participants with PDA
  Interventions: Drug: RO6927005; Drug: gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: RO6927005 — RO6927005 administered intravenously on Days 1, 3, and 5 of each 21-day treatment cycle (QOD x 3).
  Arms: Part A Extension Phase Group 1; Part A Extension Phase Group 2; Part A MAD Phase RO6927005 Monotherapy
Drug: RO6927005 — RO6927005 administered intravenously on Days 1, 3, and 5 of each 28-day treatment cycle (QOD x 3).
  Arms: Part B Extension Phase; Part B MAD Phase
Drug: gemcitabine — gemcitabine administered according to local label on Days 1, 8, and 15 of each 28-day cycle.
  Arms: Part B Extension Phase; Part B MAD Phase
Drug: nab-paclitaxel — nab-paclitaxel administered according to the local label on Days 1, 8, and 15 of each 28-day cycle.
  Arms: Part B Extension Phase; Part B MAD Phase

SUMMARY:
This is a first-in-human, open-label, multi-center, Phase 1 study of RO6927005. The study will establish the safety and tolerability profile of RO6927005 and will be conducted in two parts.

In Part A, the first dose escalations will be carried out using cohorts of 1 patient. Single patient cohorts will be used to investigate increasing doses until a first dose-limiting toxicity (DLT) is reached or until grade-2 related toxicity (except infusion-related reactions), whichever comes first. At least 3 patients will be enrolled in each cohort thereafter, which, if required, can be expanded with additional patients. Part B of the study will consist of a multiple ascending dose phase (multiple patients cohorts - >/= 3 patients) followed by an extension phase of RO6927005 given in combination with gemcitabine/nab-paclitaxel.

Preliminary clinical activity will be explored throughout the study. Patients will be treated until disease progression and/or lack of clinical benefit, unacceptable toxicities, withdrawal from treatment for other reasons, death, pregnancy or termination of the study by the Sponsor, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age >/= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Patients for whom no standard curable therapy exists
* Life expectancy of >/= 12 weeks
* Last dose of systemic anti-neoplastic therapy > 21 days prior to first RO6927005 infusion
* Palliative radiotherapy is allowed up to 2 weeks before the first RO6927005 infusion; palliative 8 Gy radiotherapy is allowed during therapy.
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure must have resolved to Grade </= 1, except alopecia (any grade) and Grade 2 peripheral neuropathy
* Adequate hematological, liver, and renal function
* Negative serum or urine pregnancy test within 7 days prior to study treatment in premenopausal women and women </= 2 years after menopause (menopause is defined as amenorrhea for >/= 2 years)
* Agreement to use adequate contraceptive methods per protocol
* Measurable and/or evaluable disease as per the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1) [Groups 1, 2 of Part A and Group 3 of Part B]

Inclusion Criteria Part A: MAD

* Metastatic and/or locally advanced malignant solid tumors enriched in tumor types known to be mesothelin expressing
* Archival sample or fresh biopsy or tumor effusion must be available for retrospective mesothelin analysis

Inclusion Criteria Part A: MAD and Extension Phase (Group 1 and Group 2)

* Histologically confirmed metastatic and/or advanced malignant mesothelin-positive solid tumors as determined by central pathology lab review
* Patients must be willing to provide a screening and post-dose biopsy for biomarker analysis (extension phase only)
* Mesothelin-positive refractory/recurrent solid tumors, other than malignant pleural mesothelioma (MPM) and pancreatic ductal adenocarcinoma (PDA) (Group 1 only)
* Mesothelin-positive refractory/recurrent MPM (Group 2 only)

Inclusion Criteria Part B

* Histologically confirmed metastatic and/or advanced mesothelin-positive PDA as determined by central pathology lab review
* In the extension phase, patients must be willing to provide a screening and post-dose biopsy for biomarker analysis

Exclusion Criteria:

* Known or clinically suspected central nervous system (CNS) primary tumors or metastases including leptomeningeal metastases; history or clinical evidence of CNS metastases unless they have been previously treated, are asymptomatic, and have had no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days
* Evidence of significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results, including significant pulmonary disease other than primary cancer, uncontrolled diabetes mellitus, and/or significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, unstable angina, or clinically significant pericardial effusion)
* Active or uncontrolled infections
* Known HIV or known active HBV or HCV infection
* Patients with extrapleural pneumonectomy (EPP)
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
* Major surgery or significant traumatic injury < 28 days prior to the first RO6927005 infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment
* Dementia or altered mental status that would prohibit informed consent
* Live attenuated vaccinations 14 days prior to treatment
* Pregnant or breast-feeding women
* Known hypersensitivity to any of the components of RO6927005
* High doses of systemic corticosteroids within 7 days prior to first dosing. High dose is considered as > 20 mg of dexamethasone a day (or equivalent) for > 7 consecutive days

Exclusion Criteria (Part B):

* Patients with contra-indication and/or history of severe hypersensitivity reactions to gemcitabine and/or nab-paclitaxel as mentioned in the locally approved label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of dose-limiting toxicities, adverse events, laboratory abnormalities; incidence of anti-drug antibodies, abnormal findings on physical examination, infusion-related reactions (composite outcome measure) | Until disease progression, unacceptable toxicities, withdrawal for other reasons, death, or termination of the study by the Sponsor, whichever comes first, up to 2 years 8 months

SECONDARY OUTCOMES:
Pharmacokinetic profile of RO6927005 monotherapy based on free and total plasma RO6927005 concentrations over time (area under the curve) | Up to 2 years 8 months
Pharmacokinetic profile of RO6927005 in combination with gemcitabine/nab-paclitaxel, based on free and total plasma RO6927005 concentrations over time (area under the curve) | Up to 2 years 8 months
Efficacy: objective response rate, disease control rate, duration of response, progression-free survival, overall survival (composite outcome measure) | Up to 2 years 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Bethesda, Maryland, United States
- Toronto, Ontario, Canada
- København Ø, Denmark
- France (3):
  - Bordeaux
  - Toulouse
  - Villejuif